CLINICAL TRIAL: NCT07279922
Title: The Role of Triglyceride-glucose Index as a Predictive Marker for Insulin Resistance in Pre Diabetic Chronic Kidney Disease Patients.
Brief Title: What is the Role of Triglyceride-glucose Index as a Predictive Marker for Insulin Resistance in Pre Diabetic Chronic Kidney Disease Patients?
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Osama Ahmed Abd_elsamea, Resident at internal medicine department, Assiut University
Other Study IDs: TyG-CKD
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Disease; Pre Diabetes
MeSH Terms: conditions — Renal Insufficiency, Chronic; Glucose Intolerance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Triglyceride-glucose index — Triglyceride-glucose index calculation according to TyG index=In[Triglycerides(mg/dl)×Fasting Glucose(mg/dl)/2]

SUMMARY:
The aim of this study is to evaluate the role of the triglyceride-glucose (TyG) index as a predictive marker for insulin resistance in pre-diabetic patients with chronic kidney disease (CKD), and to investigate its potential utility as a simple, non-invasive alternative to traditional insulin resistance assessment methods.

DETAILED DESCRIPTION:
Diabetes mellitus remains a major public health challenge worldwide due to its increasing prevalence and associated complications, particularly when undiagnosed in its early stages. Early identification of individuals at high risk is essential for timely intervention to delay or prevent disease onset. Traditional diagnostic tools may miss early metabolic disturbances, necessitating more sensitive and accessible biomarkers.

The triglyceride-glucose (TyG) index, derived from fasting plasma triglycerides and glucose, has recently emerged as a simple, reliable, and cost-effective surrogate marker for insulin resistance. Its utility has been validated in multiple populations, showing strong associations with metabolic dysfunction and future development of diabetes.

Renal dysfunction is frequently associated with alterations in glucose and lipid metabolism, even before overt diabetes develops. However, the diagnostic accuracy of traditional risk markers may be compromised in the context of impaired kidney function. The TyG index offers potential advantages due to its independence from insulin measurements and ease of calculation.

Despite growing evidence on the predictive role of the TyG index, limited data exist regarding its performance across different levels of kidney function. Investigating its diagnostic value in patients with and without renal impairment may provide a valuable tool for early diabetes risk assessment and targeted preventive strategies.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years

Patients with medical history free from renal dysfunction

Patients with renal dysfunction (CKD stages 2_5 based on KDIGO guidelines)

No previous diagnosis of diabetes mellitus

Provided informed consent

Exclusion Criteria:

* Known type 1 or type 2 diabetes mellitus

Acute kidney injury

Use of steroids or medications that affect glucose and lipid metabolism

Pregnancy

Active infections

Malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged ≥18 years with medical history free from renal dysfunction or with renal dysfunction (CKD stages 2_5 based on KDIGO guidelines)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of TyG index | 2 years
  Diagnostic performance of TyG index in predicting prediabetics and diabetic patients.